CLINICAL TRIAL: NCT06263023
Title: An Observational Study of a Dedicated Preservation and Assessment Service to Optimize Organ Utilization for Hard-to-Place Kidneys
Brief Title: A Central Preservation and Assessment Service to Optimize Donor Kidney Allocation
Acronym: OPTIMAL
Status: Active, not recruiting | Type: Observational
Sponsor: 34 Lives, PBC (Industry)
Collaborators: Indiana University Health (Other); University of Miami (Other); MOUNT SINAI HOSPITAL (Other); University of Wisconsin, Madison (Other); Erie County Medical Center, Buffalo, NY (Unknown); Duke University Hospital, USA (Unknown); Barnes-Jewish Hospital (Other); Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 34L-CP-02-009
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Organ Preservation
Keywords: SNMP; Preservation; Transplantation; Kidney
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sponsor will collect kidney perfusate and urine samples at 90- and 120-minutes during SNMP to store in a -80C specimen freezer for future analysis or quality assurance. Sponsor will collect a 4mm core punch biopsy at the superior pole of the kidney for research use. Research testing of samples may include cytokine, ATP, metabolomics, transcriptomics, proteomics, genomics, dynamic contrast imagery (DCI) and/or hematoxylin and eosin (H&E) histologic staining. All donor kidneys enrolled in this study will have legally authorized consent for organ donation for transplant and research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hard-to-Place (HTP) Donor Kidneys: The study will be open to all eligible HTP kidneys from male and female donors at all participating Organ Procurement Organization (OPO) study sites. Consent for both organ donation for transplant and medical research will be obtained from the legally authorized party (LAP) by the OPO Coordinator using industry standard consent procedures and documents.
  Interventions: Other: Sub-Normothermic Machine Preservation and Assessment

INTERVENTIONS:
Other: Sub-Normothermic Machine Preservation and Assessment — Human kidneys from HTP deceased donors will be transported to the Sponsor's central preservation and assessment facility and placed onto a machine perfusion system in a sterile operating room for a brief period of Sub-Normothermic Machine Perfusion (SNMP). Basic parameters including internal renal resistance, oxygen, and electrolyte levels will be recorded using standard point-of-care hospital analyzers. Accepted kidneys will be transported to a participating transplant center using a portable oxygenated LifePort Hypothermic Machine Preservation (HMP) device.

SUMMARY:
This is a study to collect information to assess if transporting hard-to-place (HTP) donor kidneys to a central preservation and assessment facility with dedicated organ assessment capabilities increases allocation success to transplant hospitals.

DETAILED DESCRIPTION:
This is an Observational study of a centralized kidney assessment facility providing brief sub-normothermic machine perfusion (SNMP) to HTP donor kidneys to provide transplant centers additional information for accepting HTP kidneys.

This study is intended to collect data to evaluate the feasibility of a dedicated central service to determine if additional assessment data helps increase allocation to transplant centers. Transplantation will follow standard-of-care at each transplant center, including required post-transplant data collection, which must be reported to the OPTN registry by the center.

ELIGIBILITY:
Donor Kidney Inclusion Criteria:

* Be considered HTP, by receiving refusals from every transplant center within the 250 nm allocation radius or similar definition by the local OPO.
* From a Male or female deceased donor, aged 16- 75 years old.
* Kidney initially procured, preserved, and packaged with intent to transplant.
* LAP provides informed consent for organ donation for transplant and research purposes.
* The HTP donor kidney must be allocated to a participating transplant center by a participating OPO, and the transplant center makes the decision to send kidney to Sponsor's central preservation and assessment facility for SNMP assessment and preservation prior to determining suitability for allocation.

Donor Kidney Exclusion Criteria:

* From a Donor with pre-admission diagnosis of end stage renal failure.
* Obvious surgical damage to artery(s), vein(s), or ureter(s) preventing machine perfusion.
* From a donor with confirmed HIV (+), HBVSAg (+) and/or HCV NAT (+) serology results.
* No LAP consent for both transplant and research purposes.
* Cannot arrive to Sponsor's central preservation and assessment facility before reaching 24 hours of cold ischemic time (CIT).

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes hard-to-place (HTP) deceased donor kidneys retrieved from donation after brain death (DBD) and donation after circulatory death (DCD) donors aged 16- 75.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Transplant Allocation Success | 1 year
  The primary objective for this study is a 50% success rate or higher for allocation of Hard-to-Place (HTP) kidneys to a participating transplant center after sNMP assessment at the Sponsor's central facility.

SECONDARY OUTCOMES:
7-Day Delayed Graft Function (DGF) | 7 days post-transplant
  Requirement for dialysis within first 7 days post-transplant
Graft Survival | 1- and 3-months post-transplant
  Donor kidney survival
Patient Survival | 1- and 3-months post-transplant
  Recipient survival
Serum Creatinine (sCr) | 1- and 3-months post-transplant
  Recipient sCr
eGFR | 1- and 3-months post-transplant
  Recipient estimated glomerular filtration rate
Long term data collection- Graft Survival | Annually, up to 3-years post-transplant
  Graft survival
Long term data collection- Patient Survival | Annually, up to 3-years post-transplant
  Patient survival
Long term data collection- Serum Creatinine | Annually, up to 3-years post-transplant
  Recipient sCr
Long term data collection- eGFR | Annually, up to 3-years post-transplant
  Recipient estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Chris Jaynes, Principal Investigator — 34 Lives, PBC (Sponsor)
Locations (8):
- United States (8):
  - Edward Hines, Jr. VA Hospital, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Erie County Medical Center, Buffalo, New York
  - New York University Langone, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Standard data will be obtained from the Organ Procurement and Transplantation Network (OPTN), which is readily available to the public via request to the Health Resources Service Administration (HRSA), in de-identified form to protect privacy. These standard data include information about the organ donor, preservation procedure, the recipient's kidney transplant, and post-operative follow-up.

REFERENCES:
- [Background] Kayler LK, Nie J, Noyes K. Hardest-to-place kidney transplant outcomes in the United States. Am J Transplant. 2021 Nov;21(11):3663-3672. doi: 10.1111/ajt.16739. Epub 2021 Jul 20. PMID 34212471
- [Background] Hosgood SA, Callaghan CJ, Wilson CH, Smith L, Mullings J, Mehew J, Oniscu GC, Phillips BL, Bates L, Nicholson ML. Normothermic machine perfusion versus static cold storage in donation after circulatory death kidney transplantation: a randomized controlled trial. Nat Med. 2023 Jun;29(6):1511-1519. doi: 10.1038/s41591-023-02376-7. Epub 2023 May 25. PMID 37231075
- [Background] Minor T, von Horn C, Gallinat A, Kaths M, Kribben A, Treckmann J, Paul A. First-in-man controlled rewarming and normothermic perfusion with cell-free solution of a kidney prior to transplantation. Am J Transplant. 2020 Apr;20(4):1192-1195. doi: 10.1111/ajt.15647. Epub 2019 Nov 10. PMID 31599063